CLINICAL TRIAL: NCT01473901
Title: A Phase I, Two-stage, Multi-center, Open Label, Dose-escalation Study of BKM120 in Combination With Adjuvant Temozolomide and With Concomitant Radiation Therapy and Temozolomide in Patients With Newly Diagnosed Glioblastoma
Brief Title: A Phase I Dose Escalation Study of BKM120 With Radiation Therapy and Temozolomide in Patients With Newly Diagnosed Glioblastoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CBKM120E2101; 2011-001157-87 (EudraCT Number)
Record Dates: First submitted 2011-08-18; First posted 2011-11-17 (Estimated); Last update posted 2020-12-09 (Actual); Status verified 2017-09

CONDITIONS: Glioblastoma
Keywords: BKM120; temozolomide; glioblastoma multiforme; GBM; Newly diagnosed
MeSH Terms: conditions — Glioblastoma | interventions — NVP-BKM120; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BKM120 + Temozolomide (Concomitant Phase) (Experimental): Cranial radiation: Days 1 - 5 every 7 days for 42 days60 Gy in 30 fractions; Temozolomide: 75 mg/m2 Daily, orally; BKM120: 0, or 40, or 60, or 80 mg/d Daily, orally or Days 1-5 every 7 days, orally
  Interventions: Drug: BKM120 + temozolomide
- BKM120 + temozolomide with/without radiotherapy (Experimental): Adjuvant phase cycle 1:
  Temozolomide 150 mg/m2 - Days 1 - 5 every 28 days Daily; BKM120 60, or 80, or 100 mg/d;
  Adjuvant phase cycle 2+:
  Temozolomide 200* mg/m2 - Day 1 ~ 5 every 28 days Daily BKM120 0, or 40, or 60, or 80 or 100 mg/d
  Interventions: Drug: BKM120 +temozolomide with/without radiotherapy

INTERVENTIONS:
Drug: BKM120 + temozolomide — The investigational drug, BKM120, will be supplied as 10-mg and 50-mg hard gelatin capsules. BKM120 will be administered on a once daily dosing schedule at a dose of 40 mg, or 60 mg, or 80 mg, or 100 mg (p.o.), in combination with the approved dosing of temozolomide and SoC delivery of cranial irradiation for GBM. The patient will be dosed with BKM120 on a flat scale of mg/day and the dose of BKM120 will not be adjusted to body weight or body surface area. Patients should not eat for 2 hours after the administration of BKM120. Temozolomide in 5 mg, 20 mg, 100 mg, 140 mg, 180 mg or 250 mg capsules will be administered in combination with the investigational drug BKM120.
  Arms: BKM120 + Temozolomide (Concomitant Phase)
Drug: BKM120 +temozolomide with/without radiotherapy — The investigational drug, BKM120, will be supplied as 10-mg and 50-mg hard gelatin capsules. BKM120 will be administered on a continuous once daily dosing schedule at a dose of 40 mg, or 60 mg, or 80 mg, or 100 mg (p.o.), in combination with the approved dosing of temozolomide and SoC delivery of cranial irradiation for GBM. The patient will be dosed with BKM120 on a flat scale of mg/day and the dose of BKM120 will not be adjusted to body weight or body surface area. Patients should not eat for 2 hours after the administration of BKM120. Temozolomide in 5 mg, 20 mg, 100 mg, 140 mg, 180 mg or 250 mg capsules will be administered in combination with the investigational drug BKM120.
  Arms: BKM120 + temozolomide with/without radiotherapy

SUMMARY:
This clinical study will assess the doses of BKM120 appropriate for patients with newly diagnosed glioblastoma when given in combination with radiotherapy and temozolomide.

ELIGIBILITY:
Inclusion Criteria:

* Patient is ≥ 18 years of age on the day of consent signature
* Patient with histologically demonstrated, previously untreated glioblastoma
* Patient may have received initial treatment for GBM as follows:

  * For patients enrolled into Stage I, they must have received at least 75% of planned radiotherapy (60 Gy) with temozolomide treatment during the concomitant phase have documentation that the patient's absolute neutrophil count (ANC) is ≥ 1.5 x 109/L, platelet count is ≥ 100 x 109/L, and there was no CTC grade 2 or above nonhematological toxicity (except for alopecia, nausea, vomiting) during the concomitant phase treatment be within ≥ 4 weeks but ≤ 6 weeks following the completion of temozolomide in the concomitant phase
  * For patients enrolled into Stage II, they must be within ≥ 2 weeks but ≤ 6 weeks after primary GBM resection/biopsy The patient must have recovered from the definitive surgical procedure for GBM
* Patient is able to be assessed by periodic dynamic contrast enhanced magnetic resonance imaging (DCE-MRI) scan
* Patient has Karnofsky performance status >= 60
* Patient has adequate bone marrow and organ function

Exclusion Criteria:

* Patient has received previous treatment with PI3K and/or mTOR inhibitors for GBM or for pre-existing neoplasm transformed to GBM. Patient has received any prior anti-neoplastic therapy for BKM, except for the treatment allowed in inclusion criteria
* Patient has any tumor progression after definitive GBM resection/ biopsy, except for the transformation from previous low grade glioma. Patient with a concurrent malignancy or malignancy within 3 years of study enrollment (with the exception of adequately treated, basal or squamous cell carcinoma, non-melanomatous skin cancer or curatively resected cervical cancer)
* Patient who had not recovered to grade 1 or better from any adverse events (except alopecia, nausea, vomiting) related to previous antineoplastic therapy before screening procedures are initiated, as allowed in inclusion criteria
* Patient has any of the following baseline mood disorders (not attributable to GBM) as judged by the Investigator or a Psychiatrist, or meets the cut-off score of ≥ 12 in the PHQ- 9 or a cut-off of ≥ 15 in the GAD-7 mood scale for reasons not attributable to GBM; or selects a positive response of '1, 2, 3' to question number 9 regarding potential for suicidal thoughts or ideation in the PHQ-9 (independent of the total score of the PHQ-9)
* Medically documented history of or active major depressive episode, bipolar disorder (I or II), obsessive-compulsive disorder, schizophrenia, a history of suicidal attempt or ideation, or homicidal ideation (immediate risk of doing harm to others)
* Active severe personality disorders (defined according to DSM-IV). Note: for patients with psychotropic treatments ongoing at baseline, the dose and the schedule should not be modified within the previous 6 weeks prior to start of study drug.
* ≥ CTCAE grade 3 anxiety
* Patient who is concurrently using any other approved or investigational anti-neoplastic agent
* Patient who has undergone the following invasive procedures: Major surgical procedure, open biopsy or significant traumatic injury < 14 days prior to starting study drug or has not recovered from side effects of such therapy, anticipation of need for invasive surgical procedure during the course of the study, biopsy within 7 days prior to starting study drug
* Patient has poorly controlled diabetes mellitus (HbA1c > 8%)
* Patient is currently receiving increasing or chronic treatment with corticosteroids or another immunosuppressive agent
* Patient is currently receiving an enzyme inducing anti-epileptic drug. The patient must have discontinued EIAED therapy for at least two weeks prior to starting study drug. Non-enzyme inducing anti-epileptic medication is allowed, except those listed in the protocol

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2011-12-30 (Actual); Primary Completion 2017-05-17 (Actual); Study Completion 2017-05-17 (Actual)

PRIMARY OUTCOMES:
Dose Limiting Toxicity (DLT) | Concomitant phase (42 days), adjuvant phase cycle 1 (28-day cycle), adjuvant phase cycles 2 (28-day cycle)
  Per DLT criteria as defined in protocol

SECONDARY OUTCOMES:
No of participants with Adverse events based on abnormal laboratory results, abnormal electrocardiogram (ECG) findings | Baseline, 30 days post the last BKM120 treatment
  Per common terminology criteria for adverse events (CTCAE) criteria (version 4.0)
Objective response rate (ORR) | Baseline, 18 months after first BKM120 treatment
  Antitumor activity will be assessed using the Neuro-Oncology Working Group updated response assessment criteria for high grade gliomas - per RANO criteria.
Progression free survival (PFS) | at 12 months and at 18 months
  Per patient survival follow up feedbacks
Overall survival (OS) | Until death or consent withdrawal
  Per patient survival follow up feedbacks
Plasma concentration-time profiles and basic pharmacokinetic parameters of BKM120 and temozolomide (Cmax, tmas, AUC, half-life) | baseline, Day 1, 8, 15, 28 in concomitant phase, Cycle 1 Day 1, 5 and Cycle 2 Day1, 5 at adjuvant phase (28-day per cycle)
  Standard bioanalytical-pharmacokinetic (PK) analysis on PK samples for BKM120 and temozolomide.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (8):
- United States (3):
  - Highlands Oncology Group Highlands Oncology, Fayetteville, Arkansas
  - Dana Farber Cancer Institute SC (1), Boston, Massachusetts
  - University of Texas/MD Anderson Cancer Center MD Anderson DeGrout, Houston, Texas
- Novartis Investigative Site, Melbourne, Victoria, Australia
- Canada (2):
  - Novartis Investigative Site, Hamilton, Ontario
  - Novartis Investigative Site, Toronto, Ontario
- Spain (2):
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Madrid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wen PY, Rodon JA, Mason W, Beck JT, DeGroot J, Donnet V, Mills D, El-Hashimy M, Rosenthal M. Phase I, open-label, multicentre study of buparlisib in combination with temozolomide or with concomitant radiation therapy and temozolomide in patients with newly diagnosed glioblastoma. ESMO Open. 2020 Jul;5(4):e000673. doi: 10.1136/esmoopen-2020-000673. PMID 32661186
- See also: Results for CBKM120E2101 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=17131